CLINICAL TRIAL: NCT04351607
Title: Einfluss Eines Oralen Eisenpräparats Mit Hoher Bioverfügbarkeit (OLEOvital® EISEN FORTE) Auf Die präoperative Hämoglobinkonzentration Bei anämischen Patienten
Brief Title: Preoperative Supplementation of Sucrosomal Iron as Hematopoietic Support.
Acronym: Preop Iron
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mein Hanusch-Krankenhaus (Other)
Responsible Party: Principal Investigator, Alexander Löckinger MD., Msc., M.D. MSc., Mein Hanusch-Krankenhaus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020001
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Anemia, Iron-Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Verum (Experimental): oral dose of 2 x 30mg (=60mg) Oleovital® Eisen Forte p.o. per day over a limited intake of 3-6 weeks due to increased physiological iron demand
  Interventions: Dietary Supplement: Oleovital® Eisen Forte
- Control group (No Intervention): no intervention
- Patient with menstral bleeding - subcollective A (Other): verum or control
  Interventions: Dietary Supplement: Oleovital® Eisen Forte
- Patient without menstral bleeding - subcollective B (Other): verum or control
  Interventions: Dietary Supplement: Oleovital® Eisen Forte

INTERVENTIONS:
Dietary Supplement: Oleovital® Eisen Forte — 60 mg daily oral Supplementation for 3 to 6 weeks
  Other Names: Verum
  Arms: Patient with menstral bleeding - subcollective A; Patient without menstral bleeding - subcollective B; Verum

SUMMARY:
To prove, if preoperative elective anemic patients improve their hemoglobin levels within 3-6 weeks preoperativly after daily oral dietary supplementation of 60mg sucrosomal iron.

DETAILED DESCRIPTION:
Patients with preoperative anemia have a poorer perioperative outcome in morbidity and mortality as part of surgery. Oral iron preparations have so far had poor bioavailability (approx. 30%) and mostly gastrointestinal side effects that often lead to discontinuation of treatment. Intravenous iron preparations also have an increased risk of allergic disease, which has already led to deaths in Austria. Oleovital® Eisen Forte shows improved bioavailability and hardly any gastrointestinal side effects. It should be improved in anemic patients by oleovital iron forte the hemoglobin content of the blood before surgery. Preoperative anemia is a relatively common problem that has not been preoperatively treated so far and therefore studies such as the one present here are very relevant.

The dietary supplement (Oleovital® Eisen Forte) has been on the market in Austria for iron substitution since autumn 2016. Oleovital® Eisen Forte seems suitable to produce a physiological hemoglobin content. The improved galenics is without previously known gastrointestinal side effects and should be investigated in an oral dose of 2 x 30mg (=60mg) p.o. per day over a limited intake of 3-6 weeks due to increased physiological iron demand.

The main objective of the study following a confirmant approach is to verify whether a sufficiently high number of anemic patients benefit from the oral intake of a high bioavailability iron preparation (Oleovital® Eisen Forte) in the last three to six weeks before an elective intervention (profit = response = increase in hemoglobin concentration by at least 1g/dl).

This controlled, randomized, open, prospective, monocentric study (two-armed parallel group design) should be classified as a food study (application of the commercial dietary supplement Oleovital® Eisen Forte) in an interventional setting - study-specific measures: additional blood tests and intake of Oleovital® Eisen Forte, in certain cases additional for a study-specific blood test are re-quired.

There are two study arms or groups:

* Group V = Verumgroup with iron supplementation by Oleovital® Eisen Forte
* Group K = Control group without iron supplementation - This group receives the usual treatment in the hospital.

Furthermore, stratification is carried out according to the sub-collectives

* "Patients without menstrual bleeding" (subcollective A) and
* "Patients with menstrual bleeding" (subcollective B)

ELIGIBILITY:
Inclusion Criteria:

* Written consent according to previous written and oral clarification
* Elective intervention in 3-6 weeks
* Hemoglobin (Hb) -12.0g/dl
* Age >18 years
* Non-cardiac surgery

Exclusion Criteria:

* Non-business capability or legal representation
* Pregnancy
* Breastfeeding period
* Chronic diarrhoea (> 4 weeks)
* Known massive absorption restriction (e.g. short bowel syndrome)
* Known or suspected fructose intolerance
* Iron accumulation disorders: hemochromatosis, hemosiderosis
* Vegan diet
* Use of a preparation to specifically increase the body's own erythrocyte or hemoglobin concentration or production (e.g. EPO preparations, erythrocyte concentrates) in the last 4 weeks
* Permanent or preoperativeblood loss (e.g. seepage bleeding)
* Intended intake/application of another iron-supplementing preparation before surgery
* Intended use of preparations to specifically increase the body's own erythrocyte or hemoglobin concentration or production (e.g. EPO preparations, erythrocyte concentrates) prior to surgery
* Simultaneous participation in another clinical trial with insurance cover
* Foreseeable compliance issues
* Existing refractory disorder of the bone marrow: myelodysplasia
* In the case of conspicuous base laboratory towards undiagnosed hemochromatosis: increased plasma iron, increased serum ferritin and increased transferrin saturation without increased signs of inflammation (CRP), the patient is assigned to the hematological department of the Hanusch Hospital for further diagnosis.
* Acutely therapeutic anemia Hb x 8 g/dl (indication for a mandatory correction of the Hb to a clinically safe or non-therapeutic value - no randomization into the control group makes sense)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — with or without menstral bleeding
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
hemoglobin | 3 - 6 weeks
  1 g/dl increase

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anestesiology and Critical Care Medicine, Vienna, Penzing, Austria

IPD SHARING:
Plan to Share IPD: No